CLINICAL TRIAL: NCT03640182
Title: Promotion Project of Health Management Model for Chinese Medical Preventive Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other); Tri-Service General Hospital (Other); Taiwan Society of Health Promotion (Unknown); National Research Institute of Chinese Medicine, Ministry of Health and Welfare (Other Government); National Yang Ming Chiao Tung University (Other); University of Taipei (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yi-Chang Su, Professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMUH107-REC1-008
Record Dates: First submitted 2018-07-20; First posted 2018-08-21 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Preventive Medicine; Health Promotion
Keywords: Health Management Model; Chinese Medicine; Preventive Medicine; Body Constitution; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Management of TCM preventive medicine (Experimental): The Health management model include: (1) Body constitution measurement (2) Health promotion literacy education lectures (3) Medical Ba-Duan-Jin duo-in qigong practice.
  Interventions: Other: Health management model of TCM preventive medicine

INTERVENTIONS:
Other: Health management model of TCM preventive medicine — The Health management model include: (1) Body constitution measurement (2) Health promotion literacy education lectures (3) Medical Ba-Duan-Jin duo-in qigong practice.

SUMMARY:
The purpose of this project is to design a health management model of traditional Chinese medicine (TCM) preventive medicine that meets the need of healthy or suboptimal healthy people and bring up concrete policy and implementation recommendations of "promoting the development of TCM preventive medicine and health promotion services." This project will try to practice "Health management model of TCM preventive medicine" together with health promotion groups related to Taiwan Society of Health Promotion in the district of Shilin, Zhongzheng, Beitou, and Songshan in Taipei city, and plan to recruit 200 people in this promotion project.

DETAILED DESCRIPTION:
As population aging and fast-paced lifestyle go on, chronic diseases increase rapidly and preventive medicine has become the key point of science in modern days. In addition, World Health Assembly urged member states to appropriately integrate traditional and complementary medicine into health services according to the resolutions of sixty-ninth World Health Assembly.（WHA69.24）. To strengthen the foresight of health and welfare governance, Ministry of Health and Welfare lay down "2025 White Paper on Health and Welfare Policy", looking on ahead the needs of health care, preventive care, health promotion and social welfare.

With regard to "Developing traditional Chinese medicine (TCM) Health Care", the goal of "Promoting the development of TCM health promotion service" was set and the strategy of "Promoting the development of TCM preventive medicine and health promotion services" was used to develop TCM preventive medicine, which is applied to preventing disease and improving physical fitness. By establishing the TCM health care prototype of "health promotion" and "preventive medicine," this project will push the systemic development of TCM preventive medicine forward and improve suboptimal health by early intervention, proving people with multiple model choices in self-health management. This project will first form a multidisciplinary team to gather and analyze the domestic and international health promotion and management models of TCM or traditional medicine. Then systematically arrange and induct the literature references to establish the outline and draft of "Health management model of TCM preventive medicine." Furthermore, this project will try to practice "Health management model of TCM preventive medicine" together with health promotion groups related to Taiwan Society of Health Promotion in the district of Shilin, Zhongzheng, Beitou, and Songshan in Taipei city, and plan to recruit 200 people in this promotion project. The purpose of this project is to design a health management model of TCM preventive medicine that meets the need of healthy or suboptimal healthy people and bring up concrete policy and implementation recommendations of "promoting the development of TCM preventive medicine and health promotion services."

ELIGIBILITY:
Inclusion Criteria:

* more than 20 y/o.
* can walk independently, without disability
* can communicate with Chinese or Taiwanese, and understand the purpose of the study

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-09-03 (Estimated); Study Completion 2018-09-08 (Estimated)

PRIMARY OUTCOMES:
Body Constitution Scores (measured by Body Constitution Questionnaire, BCQ) | Change from Baseline Body Constitution Yang- deficiency, Yin- deficiency and Stasis Scores at 8 week
  The measurement of Body Constitution Questionnaire will come out 3 scores:
  Scores of Yang-deficiency: ranged from 19-95 Score of Yin- deficiency: ranged from 19-95 Score of Stasis: ranged from 16-80 The higher the score, the worse the Yang- deficiency, Ying- deficiency and Stasis.
  BCQ measure
Blood pressure | Change from baseline of both systolic and diastolic pressure at 8 week
  Change of both systolic and diastolic pressure after 8 week
heart rate | Change from Baseline Heart rate at 8 week
  Change of heart rate after 8 week
Heart rate variability | Change from Baseline Heart rate variability at 8 week
  Change of Heart rate variability after 8 week
Blood oxygen concentration | Change from Baseline Blood oxygen concentration at 8 week
  Change of Blood oxygen concentration after 8 week
Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline global score of Pittsburgh Sleep Quality Index at 8 week
  Change of the global score of Pittsburgh Sleep Quality Index after 8 week The higher the global score, the worse the sleep quality. If the global <=5, defined to have good sleep quality; If the global > 5, defined to have bad sleep quality.
Brief Symptom Rating Scale（BSRS-5） | Change from Baseline score of Brief Symptom Rating Scale at 8 week
  Change of the total score of the Brief Symptom Rating Scale after 8 week. Score ranged from 0-24: the higher the score the worse the physical and mental condition.
Dietary behavior Instrument | Change from Baseline score of the Dietary behavior Instrument at 8 week
  Change of total score of the Dietary behavior Instrument after 8 week. Score ranged from 0-36: the higher the score, the better the eating behavior.
Pressure index | Change from Baseline score of Pressure index at 8 week
  Change of the pressure feeling after 8 week. Score ranged from 0-12: the higher the score, the heavy the pressure feeling.
2.44 meter stand-up test | Change from Baseline 2.44 meter stand-up test at 8 week
  Change of the stand-up and walking ability after 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chang Su, PhD, Principal Investigator — China Medical University, China
Locations (1):
- Taiwan Society of Health Promotion, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No